CLINICAL TRIAL: NCT00121173
Title: A Phase I/II Clinical Trial of pNGVL4a-Sig/E7 (Detox)/HSP70 for the Treatment of Patients With HPV 16+ Cervical Intraepithelial Neoplasia 2/3 (CIN2/3)
Brief Title: Vaccine Therapy in Preventing Cervical Cancer in Patients With Cervical Intraepithelial Neoplasia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: J0323 CDR0000439494; R21CA105696 (NIH); P30CA006973 (NIH); JHOC-J0323; JHOC-03-05-06-02 (Other: JHM IRB)
Record Dates: First submitted 2005-07-19; First posted 2005-07-21 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-06

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental): 3-500mcg doses of pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine administered IM at one month intervals.
  Genetic (recombinant DNA vaccine)
  Interventions: Biological: pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine
- Intermediate dose (Experimental): 3-1mg doses of pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine administered IM at one month intervals Genetic (recombinant DNA vaccine)
  Interventions: Biological: pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine
- High dose (Experimental): 3-3mg doses of pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine administered IM at one month intervals Genetic (recombinant DNA vaccine)
  Interventions: Biological: pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine

INTERVENTIONS:
Biological: pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine — recombinant DNA vaccine

SUMMARY:
RATIONALE: Vaccines made from protein and DNA may help the body build an effective immune response to kill abnormal cells in the cervix. The use of vaccine therapy may prevent cervical cancer.

PURPOSE: This phase I/II trial is studying the side effects and best dose of vaccine therapy and to see how well it works in preventing cervical cancer in patients with cervical intraepithelial neoplasia and human papillomavirus.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility and toxicity of pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine in preventing cervical cancer in patients with human papillomavirus (HPV)-16-positive grade 2 or 3 cervical intraepithelial neoplasia.
* Determine the effect of this vaccine on the histology of cervical tissue specimens from these patients.

Secondary

* Determine changes in lesion size and HPV viral load in patients treated with this vaccine.
* Determine the cellular, humoral, and local tissue immune responses in patients treated with this vaccine.
* Correlate measures of immune response with clinical response in patients treated with this vaccine.
* Correlate measures of immune response in patients treated with this vaccine with those observed in the preclinical model.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

* Phase I: Patients receive pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine subcutaneously once in weeks 0, 4, and 8 in the absence of disease progression or unacceptable toxicity. Patients undergo colposcopy in week 8, 15 and 19 and a therapeutic loop electrosurgical excision procedure (LEEP) in week 15.

Cohorts of patients receive escalating doses of vaccine until the safest dose is determined.

* Phase II: Patients receive vaccine as in phase I but at the safest dose determined in phase I. Patients also undergo colposcopy and LEEP as in phase I.

After completion of the study treatment, patients are followed annually for 15 years.

PROJECTED ACCRUAL: Approximately 150 patients (approximately 12 will be treated in phase I and 25 will be treated in phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cervical intraepithelial neoplasia (CIN2/3)
* Human papillomavirus-16-positive disease

PATIENT CHARACTERISTICS:

- Age: > 18

Other

* Not pregnant
* Immunocompetent

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L. Trimble, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Trimble CL, Peng S, Kos F, Gravitt P, Viscidi R, Sugar E, Pardoll D, Wu TC. A phase I trial of a human papillomavirus DNA vaccine for HPV16+ cervical intraepithelial neoplasia 2/3. Clin Cancer Res. 2009 Jan 1;15(1):361-7. doi: 10.1158/1078-0432.CCR-08-1725. PMID 19118066

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose: 3-500mcg doses of pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine administered IM
  pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine
- Intermediate Dose: 3-1mg doses of pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine administered IM
  pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine
- High Dose: 3-3mg doses of pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine administered IM
  pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine
Period: Overall Study
Arm/Group | Low Dose | Intermediate Dose | High Dose
Started | 4 | 3 | 9
Completed | 3 | 3 | 9
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | Intermediate Dose | High Dose | Total
Number analyzed (Participants) | 3 | 3 | 9 | 15
Age, Categorical [Count of Participants; unit: Participants] — Participants age 18 and older
  Participants
    <=18 years | 1 | 0 | 0 | 1
    Between 18 and 65 years | 2 | 3 | 9 | 14
    >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] — Participants ages 18 and older
  years | 26 [18 to 36] | 29 [20 to 46] | 30.3 [20 to 45] | 28.4 [18 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 9 | 15
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 2 | 2 | 9 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 1 | 1 | 7 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Safety and Toxicity
Description: Number of participants with serious adverse events (SAE) according to CTCAE 3.0 grading.
Time Frame: for the duration of the study, and whenever possible, for an additional 5 years
Population: per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | Intermediate Dose | High Dose
Number analyzed (Participants) | 3 | 3 | 9
Participants | 0 | 0 | 0

2. Primary Outcome: Efficacy
Description: The efficacy of pNGVL4a-SigE7(detox)HSP70 DNA vaccine, administered intra-muscularly. This is reported as number of participants with histologic regression of CIN2/3 to CIN1 or less by colposcopically-directed biopsy.
Time Frame: for the duration of the study, and whenever possible, for an additional 5 years
Population: per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | Intermediate Dose | High Dose
Number analyzed (Participants) | 3 | 3 | 9
Participants | 0 | 0 | 3

3. Secondary Outcome: Regression of CIN3 Lesions
Description: Number of participants with absence of CIN3 lesions at week 15
Time Frame: 15 weeks
Population: per protocol; participants who had no CIN3 lesions assessed by colposcopy and biopsy(ies) at the week 15 visit
Measure: Count of Participants; unit: Participants
Groups:
- Low Dose: 3-500mcg doses of pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine administered IM at one month intervals.
  Genetic (recombinant DNA vaccine)
  pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine: recombinant DNA vaccine
Arm/Group | Low Dose | Intermediate Dose | High Dose
Number analyzed (Participants) | 3 | 3 | 9
Participants | 0 | 0 | 3

4. Secondary Outcome: Number of Participants With T-cell Immune Responses in the Blood
Description: Systemic T-cell response as measured by γ-INF enzyme-linked immunospot assays (ELISpot)
Time Frame: 41 weeks
Population: all patients who completed all 3 vaccinations
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | Intermediate Dose | High Dose
Number analyzed (Participants) | 3 | 3 | 9
Participants | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Correlated Measures of Immune Response With Clinical Response
Description: Number of participants whose t-cell immune responses correlated with histologic regression of disease or viral clearance of HPV
Time Frame: 9 months
Population: All participants who received all 3 vaccinations
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | Intermediate Dose | High Dose
Number analyzed (Participants) | 3 | 3 | 9
Participants | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Correlated Measures of Immune Responses With the Preclinical Model
Description: Number of participants whose T-cell immune responses correlated with the immune responses observed in the preclinical model
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | Intermediate Dose | High Dose
Number analyzed (Participants) | 3 | 3 | 9
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 19 weeks
Arm/Group | Low Dose | Intermediate Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=3) | Intermediate Dose (N=3) | High Dose (N=9)
Fatigue/tiredness, flu-like symptoms (General disorders) | 2 (2) | 1 (1) | 2 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 3 (4) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was completed, as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No